CLINICAL TRIAL: NCT00505687
Title: A Multicenter, Multinational, Phase 3b, Open-Label Extension Trial to Assess the Safety and Tolerability of Long-Term Treatment of Rotigotine Patch in Subjects With Idiopathic Parkinson's Disease
Brief Title: An Open-Label Extension Trial to Assess the Safety and Tolerability of Long Term Treatment of Rotigotine in Subjects With Idiopathic Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0833; 2004-002641-12 (EudraCT Number)
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Results first posted 2010-01-12 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2010-09

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Rotigotine; Neupro®
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rotigotine (Experimental): Rotigotine
  Interventions: Drug: Rotigotine

INTERVENTIONS:
Drug: Rotigotine — Rotigotine transdermal patches:
  10 cm2 (2 mg/24 hours); 20 cm2 (4 mg/24 hours); 30 cm2 (6 mg/24 hours); 40 cm2 (8 mg/24 hours)
  Optimal dosing:
  The maximum rotigotine dose allowed is 16 mg/24 hours.
  Other Names: Neupro

SUMMARY:
The objective of this open-label extension is to assess the safety and tolerability of long-term treatment of rotigotine in subjects with idiopathic PD.

DETAILED DESCRIPTION:
This is the open-label extension to the open-label trials SP824 (NCT00242008), SP825 (NCT00243971), and SP826 (NCT00243945) that assessed the efficacy and safety and tolerability of rotigotine in subjects with idiopathic Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed treatment in one of the SP824 (NCT00242008), SP825 (NCT00243971), or SP826 (NCT00243945) trials

Exclusion Criteria:

* Subjects who had an ongoing serious adverse event from the previous OLE trial that was assessed as related to study medication

Min Age: 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2005-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (26):
- United States (9):
  - Birmingham, Alabama
  - St. Petersburg, Florida
  - Fort Wayne, Indiana
  - Southfield, Michigan
  - Forest Hills, New York
  - Asheville, North Carolina
  - Raleigh, North Carolina
  - Houston, Texas
  - Milwaukee, Wisconsin
- Innsbruck, Austria
- Germany (4):
  - Bochum
  - Dresden
  - Kassel
  - Ulm
- Tel Aviv, Israel
- Italy (3):
  - Ancona
  - Lucca
  - Messina
- South Africa (3):
  - Pretoria, Gauteng
  - Parow, Western Cape
  - Plumstead, Western Cape
- Barcelona, Spain
- United Kingdom (4):
  - Barncose Terrace, Redruth
  - Bridgend
  - North Shields
  - Tyne and Wear

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An Open-Label Extension Trial to Assess the Safety and Tolerability of Long-term Treatment of Rotigotine in Subjects with Idiopathic Parkinson's Disease in 26 locations from February 2005 to December 2008.
Groups:
- Rotigotine: Optimal dosing for Rotigotine transdermal patches, once daily: Subjects can receive a dose up to 16 mg/24 hours.
Period: Overall Study
Arm/Group | Rotigotine
Started | 186
Completed | 91
Not Completed | 95
Not completed — Important protocol violation | 2
Not completed — Lack of Efficacy | 15
Not completed — Adverse Event | 48
Not completed — Subject withdrew consent | 15
Not completed — Lost to Follow-up | 1
Not completed — Other: Underwent Implantation Of DBS | 1
Not completed — Other: Scheduled DBS Surgery | 1
Not completed — Other: Prolonged Hospitalization | 1
Not completed — Other: Patches Would Not Stick D/T Sweat | 1
Not completed — Other: Neupro Given In Hospital | 1
Not completed — Other: Disease Progression | 1
Not completed — Other: As Per Sponsor | 8

BASELINE CHARACTERISTICS:
Arm/Group | Rotigotine
Number analyzed (Participants) | 186
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 94
  >=65 years | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 126
Region of Enrollment [Number; unit: participants]
  United States | 80
  Spain | 9
  Austria | 4
  South Africa | 22
  Israel | 20
  Germany | 22
  United Kingdom | 20
  Italy | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least One Adverse Event During This Open-label Extension Study
Description: Adverse events are any untoward medical occurrences in a subject administered study treatment, whether or not these events are related to treatment.
Time Frame: four years
Population: Of the 186 subjects who entered the study, 186 are included in this summary based on the Safety Set (SS).
Measure: Number; unit: Subjects
Arm/Group | Rotigotine
Number analyzed (Participants) | 186
Subjects | 170

2. Secondary Outcome: Number of Subjects Who Withdrew From the Trial Due to an Adverse Event
Description: as for outcome 1
Time Frame: four years
Population: Of the 186 subjects who entered the study, 186 are included in this summary based on the Safety Set (SS).
Measure: Number; unit: Subjects
Arm/Group | Rotigotine
Number analyzed (Participants) | 186
Subjects | 48

3. Secondary Outcome: Mean Epworth Sleepiness Scale Score During the Open-label Extension.
Description: The Epworth Sleepiness Scale (ESS) is a self-administered questionnaire with 8 questions. The total ESS score is the sum of 8 item-scores and can range between 0 and 24. The higher the score, the higher the person's level of daytime sleepiness.
Time Frame: Visit 6 (post year 1), Visit 10 (post year 2), Visit 14 (post year 3), End of Treatment (last study visit or early withdrawal visit)
Population: Of the 186 subjects who entered the study, 186 are included in this summary based on the Safety Set (SS). Last observation carried forward (LOCF) was utilized.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 186
Score on a scale
  Visit 6 (post year 1) (n=164) | 9.3 (5.6)
  Visit 10 (post year 2) (n=164) | 10.0 (5.9)
  Visit 14 (post year 3) (n=164) | 10.3 (6.1)
  End of Treatment (n=182) | 10.1 (5.9)

ADVERSE EVENTS:
Time Frame: up to four years
Arm/Group | Rotigotine
Serious Adverse Events (participants affected / at risk) | 45/186
Other Adverse Events (participants affected / at risk) | 136/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=186)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (2)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Cellulitis (Infections and infestations) | 2 (3)
Septic shock (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Toe deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Carcinoid tumour of the small bowel (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Parkinson's disease (Nervous system disorders) | 3 (3)
Parkinsonism (Nervous system disorders) | 2 (3)
Syncope (Nervous system disorders) | 2 (2)
Hypokinesia (Nervous system disorders) | 1 (1)
Dyskinesia (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1)
Abnormal behaviour (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Urge incontinence (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Rehabilitation therapy (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=186)
Nausea (Gastrointestinal disorders) | 21 (27)
Constipation (Gastrointestinal disorders) | 12 (14)
Oedema peripheral (General disorders) | 36 (45)
Application site erythema (General disorders) | 24 (26)
Application site pruritus (General disorders) | 16 (17)
Fatigue (General disorders) | 10 (11)
Fall (Injury, poisoning and procedural complications) | 29 (47)
Back pain (Musculoskeletal and connective tissue disorders) | 21 (24)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (16)
Somnolence (Nervous system disorders) | 52 (58)
Dizziness (Nervous system disorders) | 18 (19)
Parkinson's disease (Nervous system disorders) | 10 (13)
Insomnia (Psychiatric disorders) | 24 (25)
Depression (Psychiatric disorders) | 19 (20)
Anxiety (Psychiatric disorders) | 16 (20)
Hallucination (Psychiatric disorders) | 11 (13)
Abnormal dreams (Psychiatric disorders) | 11 (11)
Sleep disorder (Psychiatric disorders) | 10 (10)
Hypertension (Vascular disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.